CLINICAL TRIAL: NCT02932436
Title: A Phase IV, Single-center, Randomized, Double-blind, Placebo-controlled, Parallel Group Study on the Effects of Empagliflozin on Left Ventricular Diastolic Function Compared to Usual Care in Individuals With Type 2 Diabetes
Brief Title: Effects of Empagliflozin on Left Ventricular Diastolic Function Compared to Usual Care in Type 2 Diabetics
Acronym: EmDia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Philipp Wild, MD, MSc, principal investigator, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UMCM-2016EPI05; 2016-001264-11 (EudraCT Number)
Record Dates: First submitted 2016-10-12; First posted 2016-10-13 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Diabetes Mellitus, Type 2; Diastolic Dysfunction
Keywords: empagliflozin; diastolic function; poorly controlled type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Empagliflozin (Experimental): 10 mg Empagliflozin daily per os for 12 weeks
  Interventions: Drug: Empagliflozin
- Placebo (Experimental): amount of Placebo corresponding to empagliflozin 10 mg daily per os for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin — 10 mg per os daily for 12 weeks
  Other Names: Jardiance
  Arms: Empagliflozin
Drug: Placebo — amount of Placebo corresponding to empagliflozin 10 mg per os daily for 12 weeks
  Arms: Placebo

SUMMARY:
The purpose of the EmDia trial is to compare the effects of empagliflozin with placebo in addition to standard diabetic treatment or dietetic treatment on cardiac diastolic function in patients with type 2 Diabetes mellitus.

DETAILED DESCRIPTION:
Diabetes is a serious and increasing global health burden. It has been shown, that diabetes is associated with a two-fold higher risk for coronary heart disease, stroke and for the aggregate of other vascular death independently of other conventional risk factors. It is the leading cause of cardiovascular disease.

Diabetes mellitus substantially increases the risk of macrovascular and microvascular complications, such as vascular dysfunction with developing coronary, cerebrovascular, and peripheral arterial disease, heart failure, nerve disorders (neuropathy), eye complications (e.g. cataracts, glaucoma diabetic retinopathy), kidney disease (nephropathy), foot ulcers, restriction of mental function, and psychosomatic diseases (e.g. stress, anxiety and depression).

The most common of the cardiovascular complications in diabetics are ischemic cardiomyopathy and left ventricular (LV) dysfunction. Of particular interest here is the diastolic dysfunction, as an early sign of diabetic heart muscle disease followed by systolic damage.

Although diabetes has a decisive role in the development of cardiovascular disease, traditional glucose lowering agents have failed to convincingly show that intensive glucose control significantly reduces CVD events.

A new approach for treatment of adult patients with type 2 diabetes was found with the selective inhibition of sodium glucose cotransporter 2 (SGLT2). Studies have shown that empagliflozin, a potent SGLT2 inhibitor, not only effectively reduces the rates of hyperglycemia but also blood pressure and weight. (16, 18) In addition, beneficial effects on arterial stiffness and vascular resistance, visceral adiposity, albuminuria and plasma urate have been reported.

The results of the EMPA-REG OUTCOME study suggest that empagliflozin added to the standard therapy has a positive influence on cardiovascular outcomes and heart failure hospitalization in individuals with diabetic mellitus.

The aim of the present study is to investigate the effects of empagliflozin, in comparison with placebo, on cardiac and vascular function as well as on cardiac biomarker in individuals with type 2 diabetes with standard therapy, increased E/E' ratio and poor glycemic control.

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting all of the following criteria at visit 0 (screening) will be considered for admission to the trial:

* Diagnosis of type 2-diabetes mellitus with stable glucose-lowering background therapy and/or dietetic treatment for at least 12 weeks
* In subjects without glucose-lowering background therapy: the application of Metformin was considered to be unsuitable due to drug intolerance
* HbA1c level of ≥6.5% and ≤10.0% at visit 0 (screening) for subjects on antidiabetic background therapy or HbA1c level of ≥6.5% and ≤9.0% for drug-naïve subjects with dietetic treatment
* Diastolic cardiac dysfunction E/E' ratio ≥8 (2D-echocardiography)
* Age 18 - 84 years
* BMI ≤ 45 kg/m² (Body Mass Index)
* For women: post-menopausal for more than 12 months without an alternative medical cause can participate in the trial. Women with childbearing potential can only participate, if they are surgically sterile or a negative pregnancy test (serum or urine) is available at visit 1 and they are willing to practice highly effective birth control method during trial. Reliable highly effective contraception comprises

  * combined (estrogen and progesteron containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal)
  * progesteron-only hormonal contraception associated with inhibition of ovaluation (oral, injectable, implantable)
  * intrauterine device (IUD)
  * intrauterine hormone-releasing system (IUS)
  * bilateral tubal occlusion
  * vasectomised partner (provided that partner is the sole sexual partner and that the vasectomised partner has received medical assessment of the surgical success)
  * sexual abstinence (defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatment. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject.
* Ability of subject to understand nature, importance and individual consequences of clinical trial
* Signed and dated informed consent of the subject must be available before start of any specific trial procedures which is consistent with ICH-GCP guidelines and local legislation

Exclusion Criteria:

Subjects presenting with any of the following criteria at visit 0 (screening) will not be included in the trial:

* Pretreatment with empagliflozin or other SGLT2 inhibitor within the last 3 months
* Pretreatment with known inducers of UGT enzymes
* Uncontrolled hyperglycemia with a glucose level > 240 mg/dl (>13.3 mmol/L) after an overnight fast
* Impaired renal function, defined as eGFR <45 ml/min/1.73 m² of body-surface-area
* End-stage renal failure or dialysis
* Severe hepatic dysfunction, defined by serum levels of either SGPT, SGOT, or alkaline phosphatase above 3 x upper limit of normal (ULN)
* Acute urinary tract infection (UTI)
* Known acute genital infection (GI)
* Symptomatic hypotension
* Hematocrit above the upper limit of the reference range
* Hypoglycemic tendencies
* Severe PAD (Fontaine classification Stage IIb - IV)
* Medical history of cancer and/or treatment for cancer within the last 5 years, subjects basalioma can be included in the study
* Medical history of pancreatitis or surgery on pancreas
* Known ketoacidosis (in the past)
* Acute febrile disease
* NYHA classification III - IV
* Pregnant and/or nursing women at visit 1 (baseline)
* Acute coronary syndrome, stroke or TIA within the last 2 months
* Planned cardiac surgery or angioplasty within 3 months
* Gastrointestinal surgeries that induce chronic malabsorption
* Blood dyscrasia or any disorders causing hemolysis or unstable Red Blood Cells (e.g. malaria, babesiosis, hemolytic anemia)
* History of hypersensitivity to the investigational medicinal product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal product
* Alcohol or drug abuse within the last 3 months that would interfere with trial participation
* Medical or psychological conditions that would jeopardize an adequate and orderly completion of the trial (at visit 0 (screening) or at visit 1 (baseline))
* Medical condition that does not allow enrollment in the trial at visit 1 (baseline)
* Current treatment with systemic steroids or change in dosage of thyroid hormones within the last 6 weeks or any other uncontrolled endocrine disorder except type 2 diabetes mellitus
* Hereditary glucose intolerance, galactose intolerance, Lapp-lactase deficiency or glucose-galactose-malabsorption
* Intake of an investigational drug in another trial within 30 days prior to intake of study medication in this trial or participating in another trial (involving an investigational drug and/or follow-up)

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2016-10-10 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
difference in E/E' ratio between 12 weeks after baseline and at baseline | 12 weeks
  difference in E/E' ratio (noninvasive surrogate marker for left ventricular diastolic function (LVEDP) measured by 2D-echocardiography) between 12 weeks after baseline and at baseline

SECONDARY OUTCOMES:
difference in E/E' ratio (change from baseline (V1) to 1 week follow-up) | 1 week
  difference in E/E' ratio (change from baseline (V1) to 1 week follow-up (2D-echocardiography)
difference in Left ventricular systolic function (LVEF) | 1 week
  difference in Left ventricular systolic function (LVEF) from baseline to week 1
difference in Left ventricular systolic function (LVEF) | 12 weeks
  difference in Left ventricular systolic function (LVEF) from baseline to week 12
difference in Left end-diastolic volume (LEDV) | 1 week
  difference in Left end-diastolic volume (LEDV) from baseline to week 1
difference in Left end-diastolic volume (LEDV) | 12 weeks
  difference in Left end-diastolic volume (LEDV) from baseline to week 12
difference in Carotid-femoral pulse wave velocity | 1 week
  difference in Carotid-femoral pulse wave velocity (cf-PWV, vascular explorer - calculated) from baseline to week 1
difference in Carotid-femoral pulse wave velocity | 12 weeks
  difference in Carotid-femoral pulse wave velocity (cf-PWV, vascular explorer - calculated) from baseline to week 12
difference in Augmentation index (AIx) | 1 week
  difference in Augmentation index (AIx, vascular explorer) from baseline to week 1
difference in Augmentation index (AIx) | 12 week
  difference in Augmentation index (AIx, vascular explorer) from baseline to week 12
difference in Arterial stiffness index (SI) | 1 week
  difference in Arterial stiffness index (SI, photo plethysmography) from baseline to week 1
difference in Arterial stiffness index (SI) | 12 weeks
  difference in Arterial stiffness index (SI, photo plethysmography) from baseline to week 12
difference in Reflection index | 1 week
  difference in Reflection index (photo plethysmography) from baseline to week 1
difference in Reflection index | 12 weeks
  difference in Reflection index (photo plethysmography) from baseline to week 12
difference in Brain natriuretic peptide (BNP) | 1 week
  difference in Brain natriuretic peptide (BNP) from baseline to week 1
difference in Brain natriuretic peptide (BNP) | 12 weeks
  difference in Brain natriuretic peptide (BNP) from baseline to week 12
difference in High sensitive troponin I (hs TnI) | 1 week
  difference in High sensitive troponin I (hs TnI) from baseline to week 1
difference in High sensitive troponin I (hs TnI) | 12 weeks
  difference in High sensitive troponin I (hs TnI) from baseline to week 12
difference in High sensitive C-reactive protein (hs CRP) | 1 week
  difference in High sensitive C-reactive protein (hs CRP) from baseline to week 1
difference in High sensitive C-reactive protein (hs CRP) | 12 weeks
  difference in High sensitive C-reactive protein (hs CRP) from baseline to week 12
difference in E/E' ratio (change from baseline (V1) to 12 weeks follow-up) in the subgroup of patients with eGFR 45-59 ml/min/1.73 m² | 12 weeks
  difference in E/E' ratio (noninvasive surrogate marker for left ventricular diastolic function (LVEDP) measured by 2D-echocardiography) between 12 weeks after baseline and at baseline in the subgroup of patients with eGFR 45-59 ml/min/1.73 m²
difference in E/E' ratio (change from baseline (V1) to 12 weeks follow-up) in the subgroup of patients with HbA1c 6.5%-6.9% | 12 weeks
  difference in E/E' ratio (noninvasive surrogate marker for left ventricular diastolic function (LVEDP) measured by 2D-echocardiography) between 12 weeks after baseline and at baseline in the subgroup of patients with with HbA1c 6.5%-6.9%

OTHER OUTCOMES:
difference in biomarkers of cardiac diseases | 1 week
  changes between baseline and follow-up after 1 week in biomarkers of cardiac diseases
difference in biomarkers of cardiac diseases | 12 weeks
  changes between baseline and follow-up after 12 weeks in biomarkers of cardiac diseases
difference in biomarkers of vascular diseases | 1 week
  changes between baseline and follow-up after 1 week in biomarkers of vascular diseases
difference in biomarkers of vascular diseases | 12 weeks
  changes between baseline and follow-up after 12 weeks in biomarkers of vascular diseases
difference in biomarkers of metabolic/diabetic status | 1 week
  changes between baseline and follow-up after 1 week in biomarkers of metabolic/diabetic status
difference in biomarkers of metabolic/diabetic status | 12 weeks
  changes between baseline and follow-up after 12 weeks in biomarkers of metabolic/diabetic status
changes in vascular/endothelial function | 1 week
  changes between baseline and follow-up after 1 week in vascular/endothelial function
changes in vascular/endothelial function | 12 weeks
  changes between baseline and follow-up after 12 weeks in vascular/endothelial function
changes in carotid atherosclerosis | 1 week
  changes between baseline and follow-up after 1 week in carotid atherosclerosis
changes in carotid atherosclerosis | 12 weeks
  changes between baseline and follow-up after 12 weeks in carotid atherosclerosis
changes in pulmonary function | 1 week
  changes between baseline and follow-up after 1 week in pulmonary function
changes in pulmonary function | 12 weeks
  changes between baseline and follow-up after 12 weeks in pulmonary function
changes in ophthalmological diseases | 1 week
  changes between baseline and follow-up after 1 week in ophthalmological diseases
changes in ophthalmological diseases | 12 weeks
  changes between baseline and follow-up after 12 weeks in ophthalmological diseases
changes in psychosomatic diseases | 1 week
  changes between baseline and follow-up after 1 week in psychosomatic diseases
changes in psychosomatic diseases | 12 weeks
  changes between baseline and follow-up after 12 weeks in psychosomatic diseases
association analysis for selected SNPs | baseline
  association analysis for selected SNPs (measured at baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Wild, MD, MSc, Principal Investigator — Johannes Gutenberg University Mainz
Locations (1):
- Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Zentrum für Kardiologie, Präventive Kardiologie und Medizinische Prävention, Mainz, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bauer KI, Baker D, Lerner R, Koeck T, Buch G, Fischer Z, Martens R, Esenkova EE, Nuber M, Andrade-Navarro MA, Ten Cate V, Tenzer S, Wild PS, Bindila L, Araldi E. Effect of Empagliflozin on the plasma lipidome in patients with type 2 diabetes mellitus: results from the EmDia clinical trial. Cardiovasc Diabetol. 2025 Sep 8;24(1):359. doi: 10.1186/s12933-025-02916-0. PMID 40922034
- [Derived] Prochaska JH, Junger C, Schulz A, Arnold N, Muller F, Heidorn MW, Baumkotter R, Zahn D, Koeck T, Trobs SO, Lackner KJ, Daiber A, Binder H, Shah SJ, Gori T, Munzel T, Wild PS. Effects of empagliflozin on left ventricular diastolic function in addition to usual care in individuals with type 2 diabetes mellitus-results from the randomized, double-blind, placebo-controlled EmDia trial. Clin Res Cardiol. 2023 Jul;112(7):911-922. doi: 10.1007/s00392-023-02164-w. Epub 2023 Feb 10. PMID 36763159
- [Derived] Junger C, Prochaska JH, Gori T, Schulz A, Binder H, Daiber A, Koeck T, Rapp S, Lackner KJ, Munzel T, Wild PS. Rationale and design of the effects of EMpagliflozin on left ventricular DIAstolic function in diabetes (EmDia) study. J Cardiovasc Med (Hagerstown). 2022 Mar 1;23(3):191-197. doi: 10.2459/JCM.0000000000001267. PMID 34939776